CLINICAL TRIAL: NCT01738919
Title: Ishiguro Extension Block Technique Versus Splinting in the Treatment of Mallet Finger Fracture. A Randomized Controlled Trial.
Brief Title: Extension Block Technique Versus Splinting in Mallet Finger Fracture.
Acronym: Ishiguro
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Janni1
Record Dates: First submitted 2012-11-28; First posted 2012-11-30 (Estimated); Results first posted 2016-11-04 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-09

CONDITIONS: Mallet Finger
MeSH Terms: interventions — Conservative Treatment; Bone Wires

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non-subluxated - splinting (Active Comparator): Conservative treatment with splinting for 6 weeks.
  Interventions: Procedure: Conservative treatment with splinting for 6 weeks.
- Non-subluxated - operation (Active Comparator): Operative treatment with extension block technique
  Interventions: Procedure: Operative treatment with extension block technique

INTERVENTIONS:
Procedure: Conservative treatment with splinting for 6 weeks. — Aluminum Karstam splints are used.
  Arms: Non-subluxated - splinting
Procedure: Operative treatment with extension block technique — Surgery with extension block technique. 6 weeks.
  Other Names: K-wires (ø= 1 mm) are used.
  Arms: Non-subluxated - operation

SUMMARY:
Mallet finger is an avulsion of the extensor tendon at its insertion on the base of the distal phalanx, with or without fracture.

Treatment af mallet finger fractures involving more than 1/3 of the articulating surface is controversial. There are to our knowledge no randomized controlled trials comparing splinting and surgical treatment with extension block technique.

The aim of this study is to compare splinting and surgical extension block fixation of mallet finger fractures in a randomized controlled trial.Our hypothesis is that conservative treatment with splinting is comparable to surgical treatment concerning functional outcome, and may even reduce the complication rates.

The original protocol was designed to include participants with non-subluxated and subluxated mallet finger fractures. However this study only included participants with non-subluxated fingers.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Mallet finger fractures with a >1mm displaced fragment involving one-third or more of the articular surface and/ or subluxation of the distal phalanges.
* Fractures with a delay of < 2 weeks.
* With reference to Wehbé and Schneider's established classification, fractures type IB and IC are included.

Exclusion Criteria:

* Open injuries
* Mallet finger fracture of the thumb
* Co-existing rheumatologic illness in the fingers
* No-compliance patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-04; Primary Completion 2015-05 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bo Munk, MD, Study Chair — Department of Hand Surgery, Aarhus University Hospital, Denmark
Locations (1):
- Department of Hand Surgery, Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited after referral of mallet fractures from the emergency department Aarhus University Hospital to the department of hand-surgery Aarhus Universityhospital.
Period: Overall Study
Arm/Group | Non-subluxated - Splinting | Non-subluxated - Operation
Started | 15 | 17
Completed | 14 | 14
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Immigrated | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Not treated in accordance to guidelines | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-subluxated - Splinting | Non-subluxated - Operation | Total
Number analyzed (Participants) | 15 | 17 | 32
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 30 [26 to 44] | 42 [26 to 51] | 31 [26 to 48]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 14
  Male | 10 | 8 | 18
Region of Enrollment [Number; unit: participants]
  Denmark | 15 | 17 | 32

OUTCOME MEASURES:

1. Primary Outcome: Extension Deficit in the Affected Distal Interphalangeal Joint.
Description: Extension deficit measured in degrees, using goniometer. (The lacking extension from at straight stretched finger = degrees of extension deficit)
Time Frame: 6 month
Measure: Mean (95% Confidence Interval); unit: degrees extension deficit
Arm/Group | Non-subluxated - Splinting | Non-subluxated - Operation
Number analyzed (Participants) | 14 | 14
degrees extension deficit | 12 [8 to 16] | 10 [4 to 16]

2. Secondary Outcome: Pain
Description: Pain in the affected join. Pain intensity were reported on a numeric rating scale (NRS), from 0-10, with 0 indicating no pain.
Time Frame: 6 month
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Non-subluxated - Splinting | Non-subluxated - Operation
Number analyzed (Participants) | 14 | 14
units on a scale | 1 [0 to 1] | 1.5 [1 to 2]

3. Secondary Outcome: Bump
Description: Number of participants with the presence of a bump on the fracture-site.
Time Frame: 6 month
Measure: Number; unit: participants
Arm/Group | Non-subluxated - Splinting | Non-subluxated - Operation
Number analyzed (Participants) | 14 | 14
participants | 7 | 5

4. Secondary Outcome: Complications
Description: Number of participants with nail deformities.
Time Frame: 6 month
Measure: Number; unit: participants
Arm/Group | Non-subluxated - Splinting | Non-subluxated - Operation
Number analyzed (Participants) | 14 | 14
participants | 2 | 4

5. Secondary Outcome: DASH
Description: Questionary: Disabilities of the Arm, Shoulder and Hand Danish version (qDASH). Scale range 0-100, with 0 indicating no disability.
Time Frame: 6 month
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Non-subluxated - Splinting | Non-subluxated - Operation
Number analyzed (Participants) | 14 | 14
units on a scale | 4.5 [0 to 9] | 12.6 [0 to 20.5]

6. Secondary Outcome: Flexion of the Distal Interphalangeal Joint.
Description: Flexion of the distal interphalangeal joint. Measured with goniometer.
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: degrees
Arm/Group | Non-subluxated - Splinting | Non-subluxated - Operation
Number analyzed (Participants) | 14 | 14
degrees | 65 [59 to 71] | 50 [39 to 61]

ADVERSE EVENTS:
Time Frame: 0-6 months observation after intervention
Arm/Group | Non-subluxated - Splinting | Non-subluxated - Operation
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/17
Other Adverse Events (participants affected / at risk) | 3/14 | 0/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Non-subluxated - Splinting (N=14) | Non-subluxated - Operation (N=14)
Secundary subluxation (Musculoskeletal and connective tissue disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No